CLINICAL TRIAL: NCT04191408
Title: Predictive Ability of PEEP Induced CVP Changes to Predict Volume Responsiveness in Mechanically Ventilated Patients After Major Abdominal Surgery
Brief Title: Predictive Ability of PEEP Induced Changes in CVP to Predict Volume Responsiveness in Mechanically Ventilated Patients After Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Andrej Šribar, MD, PhD, University Hospital Dubrava
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20196996
Record Dates: First submitted 2019-12-06; First posted 2019-12-09 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Surgery; Critical Illness; Cardiac Output, Low
MeSH Terms: conditions — Critical Illness; Cardiac Output, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mechanically ventilated patients after surgery (Experimental): After ICU admission the patient's hemodynamics (MAP, HR, CO, PPV) will be measured in supine position. It will be remeasured after PEEP has been increased from +5 to +15 cmH20. Then the baseline measurement will be repeated. Then passive leg raise will be performed and all the parameters will be remeasured.
  Interventions: Procedure: PEEP increase

INTERVENTIONS:
Procedure: PEEP increase — PEEP increase +5 to +15 cmH2O. PLR at 30 degrees.
  Other Names: Passive leg raise

SUMMARY:
Interventional study which will assess whether an positive end expiratory pressure induced increase of central venous pressure is a valid predictor of volume responsiveness in mechanically ventilated patients after major abdominal surgery assessed by increase of cardiac output after passive leg raise.

DETAILED DESCRIPTION:
Interventional study which will assess whether an positive end expiratory pressure induced increase of central venous pressure is a valid predictor of volume responsiveness in mechanically ventilated patients after major abdominal surgery assessed by increase of cardiac output after passive leg raise.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated and sedated patients admitted to the ICU after major abdominal surgery

Exclusion Criteria:

* Heart failure NYHA III or more
* Severe obstructive or restrictive lung disease
* Hypotension with MAP < 60 mmHg
* Tachycardia > 140 beats / min

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Stroke volume increase after passive leg raise | Within 30 seconds after PLR
  Patients who have a stroke volume (measured in ml) increase of 7% or more after passive leg raise will be considered volume responsive.
  After the patients have been stratified into volume responders and volume non-responders, sensitivity and specificity of PEEP induced increase in CVP and pulse pressure variation will be assessed and further statistical analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Šribar, MD, PhD, Principal Investigator — Anesthesiologist and Intensive care medicine specialist
Locations (1):
- University Hospital Dubrava, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
Might share anonymized measured data.

REFERENCES:
- [Result] Geerts BF, Aarts LP, Groeneveld AB, Jansen JR. Predicting cardiac output responses to passive leg raising by a PEEP-induced increase in central venous pressure, in cardiac surgery patients. Br J Anaesth. 2011 Aug;107(2):150-6. doi: 10.1093/bja/aer125. Epub 2011 May 27. PMID 21622963